CLINICAL TRIAL: NCT03307954
Title: Feasibility Study to Investigate the Potential Reduction of Bone Mineral Density Loss in Spinal Cord Injured Patients Using Ekso Therapy
Brief Title: Bone Mineral Density Ekso Therapy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH19034
Record Dates: First submitted 2017-09-21; First posted 2017-10-12 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2017-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ekso Therapy (Experimental): Up to 12 weeks of Ekso Therapy. Three sessions per week. One hour per session
  Interventions: Device: Ekso Therapy (Exoskeleton Suit)
- Control (Active Comparator): Up to 12 weeks of usual physiotherapy care. Three sessions per week. One hour per session.
  Interventions: Other: Usual Physiotherapy

INTERVENTIONS:
Device: Ekso Therapy (Exoskeleton Suit)
  Arms: Ekso Therapy
Other: Usual Physiotherapy
  Arms: Control

SUMMARY:
Spinal cord injury (SCI) leads to rapid and profound bone loss with large decreases in bone mineral density (BMD) below the level of the lesion. Decreases in BMD of ~2% per month from the lower limbs have been reported and rates of loss are maximal over the first two years. As a consequence, there is an increased risk of fragility fractures particularly of the lower limbs including an increased risk of hip fracture. Lower limb fragility fractures affect up to 35% of patients following SCI. These fractures are associated with considerable morbidity and an increase in mortality.

This single centre UK study will determine if it is feasible to carry out a randomised controlled BMD study in the acute SCI patient population. The study will compare the BMD of patients who receive Ekso Therapy (powered exoskeleton device) verse patients who receive usual physiotherapy alone (control group). It will address patient recruitment rates and reasons for withdrawal from the study and highlight any practicality issues with study conduct. It will also provide preliminary data on the effects of Ekso Therapy on BMD, biochemistry and bone turnover markers.

DETAILED DESCRIPTION:
There are an estimated 40,000 people living with a Spinal Cord Injury (SCI) in the UK alone (http://www.apparelyzed.com/statistics.html).

Spinal cord injury (SCI) leads to rapid and profound bone loss with large decreases in bone mineral density (BMD) below the level of the lesion (Frey-Rindova et al., 2000). Decreases in BMD of ~2% per month from the lower limbs have been reported and rates of loss are maximal over the first two years (Jiang et al., 2005). Bone loss is associated with increased bone resorption and remodelling imbalance which is thought to be due to the combined effects of immobility together with neurogenic effects. As a consequence, there is an increased risk of fragility fractures particularly of the lower limbs including an increased risk of hip fracture. Lower limb fragility fractures affect up to 35% of patients following SCI. These fractures are associated with considerable morbidity and an increase in mortality.

BMD is conventionally measured using dual-energy x-ray absorptiometry (DXA). This technique enables measurement of bone mineral content, projected area and areal BMD at the lumbar spine and proximal femur. DXA does not allow differentiation between cortical and trabecular bone and does not have the ability to examine microstructural change. High resolution peripheral quantitative computed tomography (HR-pQCT) is a novel technique which enables changes in trabecular and cortical microstructure to be evaluated. Using HR-pQCT it is possible to detect changes in surrogate measures of bone strength in response to loss of weight bearing activity over just 6 weeks (Kazakia et al, 2014).

To date, there is no established intervention which has been demonstrated to prevent or reverse bone loss and fractures in this clinical setting. Small studies have suggested that anti-resorptive agents including bisphosphonates (Bryson et al., 2009) and denosumab (Gifre et al., 2015) have potential to protect against bone loss following SCI. Physical therapy using vibration was ineffective (Dudley-Javoroski et al., 2015) as was an ambulation programme undertaken late in the management of SCI (Needham-Shropshire et al., 1997). Once bone loss has occurred, it appears to be at best only partially reversible on recovery of lower limb function. It has been postulated that weight-bearing activity on its own (Dionyssiotis et al., 2015) or perhaps in combination with anti-resorptive treatment has the potential to preserve or improve bone health following SCI.

In 2014, a new therapy service called 'Ekso Therapy' was introduced at the Sheffield Princess Royal Spinal Injuries Centre. Ekso is a revolutionary powered exoskeleton device, which is strapped on to patients with a SCI to enable them to stand and walk. The device is manufactured by Ekso Bionics and is CE marked. It has been reported to be a good form of exercise allowing patients to stretch, and is claimed to be beneficial for muscle strength, bone health, bowel and bladder function and circulation and has a positive psychological impact. None of these claims have been investigated or proven in large clinical trials.

This single centre UK study will therefore determine if it is feasible to carry out a randomised controlled bone study in the acute SCI patient population using the Ekso device. Investigators will compare the BMD of acute SCI patients before and after they receive a programme of Ekso Therapy alongside their usual physiotherapy and compare it to patients who receive standing therapy with usual physiotherapy alone (control group).

It will address patient recruitment rates and reasons for withdrawal from the study and highlight any practicality issues with study conduct. It will also provide preliminary data on the effects of Ekso Therapy on bone mineral density, biochemistry and bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years old inclusive
* Traumatic and non-traumatic incomplete tetraplegic or paraplegic patient following acute SCI injury
* Be able to provide written informed consent or verbal consent in the presence of an independent witness
* Stable medical condition
* Independently transfer from a wheelchair to a regular chair ideally by completing a "lift and shift" manoeuvre or a standing pivot transfer.
* Currently undertaking an active standing programme with a standing frame i.e. Oswestry Standing Frame, for longer than 15 minutes for inpatients
* Sufficient upper limb function to be able to grasp and release objects in the hands with or without use of 'Active hands'.
* Sufficient range of movement to tolerate sit to stand and normal walking.
* Sufficient upper extremity strength and sitting balance to assist with balance in standing with a frame and or crutches.
* Sufficient lower extremity bone density to stand in standing frame and walk in traditional orthotics
* Motor complete paralysis (Asia A) C7 or below
* Incomplete motor paralysis (Asia C) C2 or below
* Weigh 220 pounds (100 kilograms) or less
* Between 5'2" and 6'4" (157 to 188 cm) tall
* Standing hip width of 17.5" or less.

Exclusion Criteria:

* Aged less than 18 years old
* Lack the mental capacity to consent
* Ventilated patients
* Significant upper or lower limb contractures / spasticity
* Currently participating in another research study which may have an impact on the study or patient safety and well-being.
* Range of motion restrictions that would prevent clients from achieving a normal, reciprocal gait pattern, or would restrict clients completing normal sit-to-stand or stand-to-sit transitions
* Spinal instability
* Unresolved deep vein thrombosis (DVT)
* Decreased standing tolerance due to orthostatic hypotension
* Significant osteoporosis that prevents safe standing or may increase the risk of fracture caused by standing or walking
* Previous lower limb fractures less than 6 months ago.
* Uncontrolled spasticity
* Uncontrolled Autonomic Dysreflexia (AD)
* Insufficient upper extremity strength to assist with balance with frame or crutches
* Leg length discrepancy above recommended values. (Upper leg length discrepancy greater than half an inch (> .5") or lower leg discrepancy greater than three-quarters of an inch (>.75") )
* Skin integrity issues on contact surfaces of the device or on surfaces that would prohibit sitting
* Cognitive impairments resulting in motor planning or impulsivity concerns
* Pregnancy
* Ability to mobilise further than 10m on the parallel bars or with use of a walking aid.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Number of valid data sets | 2 years recruitment plus 3 months FU
  10 valid data sets (5 in each arm)

SECONDARY OUTCOMES:
Number of participants recruited | 2 years
  Recruitment of 20 patients over 2 years
Number of participants with treatment-related adverse events according to the study protocol | Up to 2 years plus 3 months FU
Bone Mineral Density | Week 0 and Week 12
  Measurement of spine, radius, ulna and hip BMD using DXA and tibia and radius BMD using hp-pqCT
Bone Biochemistry | Week 0 and Week 12
  Measurement of bone profile biochemistry, Vitamin D and PTH.
Bone Biomarkers | Week 0, Week 4, Week 8 and Week 12
  Measurement of P1NP and CTX

CONTACTS AND LOCATIONS:
Locations (1):
- Northern General Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No